CLINICAL TRIAL: NCT04846296
Title: The Turkish Adaptation, Validity and Reliability Study of the Quality of Life Profile for Spinal Deformities
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.04.121
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Quality of Life; Spinal Deformity; Scoliosis
Keywords: quality of life; scoliosis; spine; validation; adaptation
MeSH Terms: conditions — Scoliosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Between 10-16 years old Cobb angle 10-40 degrees Being treated with conservative treatment (brace- exercise) for scoliosis Accepted to answer the questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The QLPSD, developed in Spain, was the first questionnaire designed to evaluate HRQoL in adolescents with spinal deformities. It has shown good validity and reliability. English, French and Persian versions of the QLPSD have been developed and validated. Good reliability and ease of use are mentioned in these versions. The QLPSD was designed to examine adolescents with spinal deformities and measure the effect of orthotic and surgical treatments on QoL.
  Other Names: the Quality of Life Profile for Spinal Deformities

SUMMARY:
The purpose of this study is to translate and culturally adapt the quality of life profile for spinal deformities (QLPSD) to Turkish language and test the validity and reliability of Turkish version of QLPSD in patients with adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
The QLPSD, developed in Spain, was the first questionnaire designed to evaluate HRQoL in adolescents with spinal deformities. It contains 21 items in five dimensions: psychosocial functioning (7 items), sleep disturbances (4 items), back pain (3 items), body image (4 items), and back flexibility (3 items). Responses to items use a 5-point Likert scale. The possible score range is 21-105.

The QLPSD has shown good validity and reliability. English, French and Persian versions of the QLPSD have been developed and validated. Good reliability and ease of use are mentioned in these versions. The QLPSD was designed to examine adolescents with spinal deformities and measure the effect of orthotic and surgical treatments on QoL. This questionnaire is practical and suitable for patients with spinal deformities. As a result we choose to translate the QLPSD into Turkish as it is less costly, practical and time consuming than developing a new tool. QLPSD may be preferred during follow-up of the results of conservative and / or surgical treatments for spinal deformities.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10-16 years old
* Cobb angle 10-40 degrees
* Being treated with conservative treatment for spinal deformities
* Being accepted to answer the questionnaire

Exclusion Criteria:

* Being not accepted to answer the questionnaire
* Having any mental disorder to prevent participation the study

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Aged between 10-16years old with scoliosis who treated by conservative management.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Turkish adaptation, validity and reliability of QLPSD | 1 day
  The questionnaire contains 21 items in five dimensions:
  psychosocial functioning (7 items), sleep disturbances (4 items), back pain (3 items), body image (4 items), and back flexibility (3 items). Responses to items use a 5-point Likert scale. The possible score range is 21- 105. Higher scores indicate poorer QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Damla Korkmaz, 1, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Validation and Reability of the Quality of Life Profile for Spinal Deformities into Turkish population
Supporting Information: Study Protocol, SAP
Time Frame: 3 months
Access Criteria: after publication

REFERENCES:
- [Background] Feise RJ, Donaldson S, Crowther ER, Menke JM, Wright JG. Construction and validation of the scoliosis quality of life index in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1310-5. doi: 10.1097/01.brs.0000163885.12834.ca. PMID 15928558
- [Result] Schulte TL, Thielsch MT, Gosheger G, Boertz P, Terheyden JH, Wetterkamp M. German validation of the quality of life profile for spinal disorders (QLPSD). Eur Spine J. 2018 Jan;27(1):83-92. doi: 10.1007/s00586-017-5284-3. Epub 2017 Sep 9. PMID 28889338
- See also: Construction and validation of the scoliosis quality of life index in adolescent idiopathic scoliosis. — http://pubmed.ncbi.nlm.nih.gov/15928558/
- See also: German validation of the quality of life profile for spinal disorders (QLPSD) — http://pubmed.ncbi.nlm.nih.gov/28889338/